CLINICAL TRIAL: NCT01414335
Title: Amino Acid Composition Reduces Frequency of Common Cold. Results of a Controlled Randomized Completely Masked Trial
Brief Title: Amino Acid Composition Reduces Frequency of Common Cold. Results of a Controlled Completely Masked Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyberg Vital GmbH (Industry)
Responsible Party: Sponsor: Kyberg Vital GmbH, Sponsor: Kyberg Vital GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kyb10/09
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: to Improve the Effectiveness of a Amino Acid Dietary Supplement in Chronic Pharyngeal Infections vs Placebo
Keywords: amino acids; immune system; vitamins; chronic infection; common cold; ear; nose; throat
MeSH Terms: conditions — Persistent Infection; Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: Placebo
- amino acid composition (Active Comparator)
  Interventions: Dietary Supplement: amino acid composition

INTERVENTIONS:
Dietary Supplement: amino acid composition — one single pouch (13g) of amino acid mixture and vitamins diluted into 200 ml of still water. This solution was daily oral taken after a meal.
  Other Names: Brand name: aminoplus immun
  Arms: amino acid composition
Other: Placebo — placebo contained no amino acids and vitamins and was identical in appearance and solution properties.
  Other Names: remedy
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness of a dietary supplement with high dosage of amino acids and vitamins in the treatment of acute and chronic infection of pharyngeal area known as common cold. T

ELIGIBILITY:
Inclusion Criteria:

men and women with at least two episodes of common cold and infection of ear, nose and pharyngeal area.

Exclusion Criteria:

* people with severe infection like pneumonia, patients expecting an in-patient treatment during the trial, pregnant or breast feeding and people not able to understand the procedure of the treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
outcome of efficacy | 3 month treatment
  For each study day,participants recorded in a diary rectal temperature, symptoms of sneezing, blocked nose or streaming eyes, whether they had problems to swollow and whether they had headache or pain in arms or legs.

SECONDARY OUTCOMES:
outcome of efficacy | 3 month treatment
  Secondary outcome variables: feel the patient fit and able-bodied.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyberg Vital - Doris Meister, Oberhaching, Bavaria, Germany